CLINICAL TRIAL: NCT04048031
Title: A Randomized, Double-Blind, Placebo-Controlled Study Evaluating The Ability And Safety Of A Nutraceutical Supplement With Standardized Botanicals To Promote Hair Growth In Perimenopausal, Menopausal And Post-Menopausal Women With Self-Perceived Thinning Hair
Brief Title: Efficacy and Safety of a Nutraceutical Supplement With Standardized Botanicals in Peri-menopausal and Menopausal Women With Thinning Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ablon Skin Institute Research Center (Other)
Collaborators: Nutraceutical Wellness Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASIRC-NW-02
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2019-08

CONDITIONS: Hair Thinning
Keywords: Hair thinning; Hair Loss; Women; Perimenopausal, Menopausal and Post Menopausal Women; Nutraceutical supplement
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: This is a six (6) month double-blind, randomized, placebo-controlled study with a six (6) month open-label extension to assess the safety and efficacy of Nutrafol® Women's Balance oral supplement in improving hair growth in perimenopausal, menopausal and post-menopausal female subjects with self-perceived thinning hair. After an initial screening period to determine eligibility, subjects will be randomly assigned to one of the following treatment arms: Nutrafol® vs. Placebo for the initial 6 months of the trial. All subjects (Nutrafol® and placebo groups) will receive the active treatment (Nutrafol®) throughout the latter 6-month open-label extension/follow-up period.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind with a 6 month Open-Label Exension
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutrafol Supplement Capsules (Active Comparator): NUTRAFOL's Synergen Complex Plus® is a formulation based on a patent-pending Synergen Complex®, a combination of botanicals with potent anti-inflammatory, anti-stress adaptogenic, antioxidant, DHT-inhibiting and hormone-rebalancing properties - combined to synergistically combat the multiple underlying factors that compromise hair growth and health. Some key ingredients include Sensoril Ashwagandha, BCM-95 BioCurcumin, Saw Palmetto, EVNolMax 20% Tocotrienol/Tocopherol complex, gelatinized Maca, Astaxanthin, Bioperine (piperine), and Capsimax (capsaicin), all of which are bio-optimized and clinically tested.
  Subjects to take four (4) Nutrafol Supplement capsules by mouth daily for 180 days with a substantial meal.
  Interventions: Dietary Supplement: Nutrafol Supplement Capsules
- Placebo Capsules (Placebo Comparator): The placebo capsules contain no active ingredients. Subjects to take four (4) Placebo capsules by mouth daily for 180 days with a substantial meal.
  Interventions: Other: Placebo Capsules
- Open Label 6 month Extension (Other): During the 6 month open label extension all 70 subjects will receive NUTRAFOL's Synergen Complex Plus® which is a formulation based on a patent-pending Synergen Complex®, a combination of botanicals with potent anti-inflammatory, anti-stress adaptogenic, antioxidant, DHT-inhibiting and hormone-rebalancing properties - combined to synergistically combat the multiple underlying factors that compromise hair growth and health. Some key ingredients include Sensoril Ashwagandha, BCM-95 BioCurcumin, Saw Palmetto, EVNolMax 20% Tocotrienol/Tocopherol complex, gelatinized Maca, Astaxanthin, Bioperine (piperine), and Capsimax (capsaicin), all of which are bio-optimized and clinically tested.
  Subjects to take four (4) Nutrafol Supplement capsules by mouth daily for the six month extension with a substantial meal.
  Interventions: Dietary Supplement: Nutrafol Supplement Capsules

INTERVENTIONS:
Dietary Supplement: Nutrafol Supplement Capsules — NUTRAFOL's Synergen Complex Plus® is a formulation based on a patent-pending Synergen Complex®, a combination of botanicals with potent anti-inflammatory, anti-stress adaptogenic, antioxidant, DHT-inhibiting and hormone-rebalancing properties - combined to synergistically combat the multiple underlying factors that compromise hair growth and health. Some key ingredients include Sensoril Ashwagandha, BCM-95 BioCurcumin, Saw Palmetto, EVNolMax 20% Tocotrienol/Tocopherol complex, gelatinized Maca, Astaxanthin, Bioperine (piperine), and Capsimax (capsaicin), all of which are bio-optimized and clinically tested. The Nutafol supplement capsules are compared to the placebo capsules which contain no active ingredients. Four (4) capsules are taken by mouth once daily with a substantial meal.
  Arms: Nutrafol Supplement Capsules; Open Label 6 month Extension
Other: Placebo Capsules — The placebo capsules contain no active ingredients. Four (4) capsules are taken by mouth once daily with a substantial amount of food.
  Arms: Placebo Capsules

SUMMARY:
NUTRAFOL® Women's Balance supplement is a novel nutraceutical supplement, scientifically formulated to specifically target the multiple underlying causes of hair loss and thinning in women. NUTRAFOL® Women's Balance capsules are comprised of primary and secondary ingredients, designed to restore hair health from the inside out. In addition to the necessary vitamins, minerals, proteins to support the nutritional needs of hair, it also contains nutraceutical-grade botanical bioactives that are standardized and clinically tested. The formulation leverages the multidimensional properties of power plants, which possess a full spectrum of phytochemicals with innate capacities to work in synergy with each other to fulfill their specific therapeutic roles. Using the latest biotechnology, these ingredients are bio-optimized and standardized, extracted with patented methods that preserve their bioactive integrity and made more bio-available and bio-absorbable via specific patented technologies.

Ingestion of NUTRAFOL® Women's Balance supplement over a six (6) month period will strengthen and promote the growth of hairs in perimenopausal, menopausal, and post-menopausal female subjects with self-perceived thinning hair when compared to baseline and those using the placebo tablet, with further improvement during the subsequent six (6) month open-label extension period.

DETAILED DESCRIPTION:
NUTRAFOL® Women's Balance supplement is a novel nutraceutical supplement, scientifically formulated to specifically target the multiple underlying causes of hair loss and thinning in women. NUTRAFOL® Women's Balance capsules are comprised of primary and secondary ingredients, designed to restore hair health from the inside out. In addition to the necessary vitamins, minerals, proteins to support the nutritional needs of hair, it also contains nutraceutical-grade botanical bioactives that are standardized and clinically tested. The formulation leverages the multidimensional properties of power plants, which possess a full spectrum of phytochemicals with innate capacities to work in synergy with each other to fulfill their specific therapeutic roles. Using the latest biotechnology, these ingredients are bio-optimized and standardized, extracted with patented methods that preserve their bioactive integrity and made more bio-available and bio-absorbable via specific patented technologies.

NUTRAFOL's Synergen Complex Plus® is a formulation based on a patent-pending Synergen Complex®, a combination of botanicals with potent anti-inflammatory, anti-stress adaptogenic, antioxidant, DHT-inhibiting and hormone-rebalancing properties - combined to synergistically combat the multiple underlying factors that compromise hair growth and health. Some key ingredients include Sensoril Ashwagandha, BCM-95 BioCurcumin, Saw Palmetto, EVNolMax 20% Tocotrienol/Tocopherol complex, gelatinized Maca, Astaxanthin, Bioperine (piperine), and Capsimax (capsaicin), all of which are bio-optimized and clinically tested.

Ingestion of NUTRAFOL® Women's Balance supplement over a six (6) month period will strengthen and promote the growth of hairs in perimenopausal, menopausal, and post-menopausal female subjects with self-perceived thinning hair when compared to baseline and those using the placebo tablet, with further improvement during the subsequent six (6) month open-label extension period. The primary endpoints will be favorable analysis using the Canon Power Shot G16 with 3GEN Dermlite FOTO Pro for macrophotography hair count analysis of terminal, vellus and total hairs at three (3) and six (6) months. The secondary endpoints will include favorable analysis using the Canon Power Shot G16 with 3GEN Dermlite FOTO Pro for macrophotography hair count analysis of terminal, vellus and total hairs at nine (9) and twelve (12) month visits. Other secondary endpoints will be favorable improvement in terminal hair diameter measured by the Dino-Lite Digital Microscopic, favorable improvement in the Blinded Physician Global Hair Assessments for hair growth and hair quality, decrease in hair shed counts with Hair Washing Procedure, statistically significant positive feedback on the Women's Hair Loss Quality of Life, Self-Assessment, Subject Treatment Satisfaction and Ease of Use, Subject Hair Satisfaction and Menopause Rating Scale Questionnaires at the three (3), six (6), nine (9) and twelve (12) month visits. The exploratory endpoint would be favorable improvement in the Hair Check device hair bundle measurement for Hair Mass Index (HMI) at the three (3), six (6), nine (9) and twelve (12) month visits. See Table of Study Procedures.

A minimum of seventy (70) female subjects will be enrolled in this clinical study; Forty (40) subjects will receive active and Thirty (30) subjects will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* 1. Females, age 40-65, who are perimenopausal, menopausal or post-menopausal. Perimenopausal is defined as increased variability in menstrual cycle length and defined as persistent difference of 7 days or more in length of consecutive cycles. Later stages include amenorrhea for 60 days or longer and/or vasomotor symptoms. These should have been present for at least 6 months prior to study. Menopause is defined as absence of menstrual bleeding for at least 12 months or 12 months status post complete Hysterectomy with Oophorectomy.

  2. Clinically-determined general good health as determined by responses to the initial study assessment.

  3. Females with self-perceived thinning hair as confirmed on initial study assessment by the Investigator (This will not include patients with medically diagnosed telogen effluvium).

  4. Females willing to maintain their normal hair shampooing frequency.

  5. Females willing to add the provided oral supplement to their current daily routine.

  6. Females willing to not substantially change their current diet, medications, or exercise routines for the duration of the study. If a subject receives physician guidance during the study to change diet, medications, or exercise routine, the subject will need to notify the clinic as soon as possible.

  7. Females willing to undergo a brief physical exam to include height, weight, blood pressure, pulse, general physical findings and a scalp exam. The physical exam will occur at Visits 1, 2, 3, 4 and 5.

  8. Females with Fitzpatrick I-IV photo skin types.

  9. Willingness to have 2D digital photography of the entire head/hair region for overall evaluation of general hair growth and fullness at Visits 1, 2, 3, 4 and 5.

  10. Willingness to have digital macrophotography of the target area and scalp for hair counts at Visits 1, 2, 3, 4 and 5.

  11. Willingness to have a bundle of hair measured by the Hair Check device for Hair Mass Index (HMI) at Visits 1, 2, 3, 4 and 5.

  12. Willingness to have ten (10) terminal hairs cut at the base of the scalp from just outside the HMI measurement area for microscopic hair measurements at Visits 1, 2, 3, 4 and 5.

  13. Willingness to have their hair washed (shampooed) over a sink containing cheesecloth for hair shedding counts at Visits 1, 2, 3, 4 and 5.

  14. Willingness to maintain a consistent hair cut and hair color throughout the 12 month study period and to come to visits with clean, dry hair.

  15. Willingness of subjects who have color treated hair to have the color treatment performed at the same time interval prior to each visit (ie. If on Visit 1 the color treatment was done one week prior then the color treatment is expected to occur at a similar interval of one week prior to Visits 2, 3, 4 and 5).

  16. Willingness of subjects to answer questionnaires related to general lifestyle, quality of life related to hair loss, self-assessment, subject treatment satisfaction and ease of use, subject hair satisfaction and the menopause rating scale at Visits 1, 2, 3, 4 and 5.

Exclusion Criteria:

1. Females who are of childbearing potential defined as still having a menstrual cycle on a regular basis who are not perimenopausal, menopausal or post-menopausal.
2. Females with any known allergy or sensitivity to any shampoo/conditioner.
3. Females with known stressful incident within the last six months (ie. death in family).
4. Females who are participating on any clinical research study at ASIRC or at another research center or doctors office.
5. Females who have recently (within the last 6 months) started the use of hormone replacement therapy (HRT). Women currently using hormones for HRT must have been on a stable dose (6 months or longer) in order to be eligible for the study (the initiation of HRT should not have been associated with the initiation of hair loss/thinning).
6. Females currently using any Low Level Laser Therapy (LLLT) to treat thinning hair.
7. Females who have regularly used Rogaine (Minoxidil) within the last 3 months.
8. Females who have used prescription drugs known to affect the hair growth cycle within the last 6 months (e.g., cyproterone acetate, aldactone/spironolactone, Finasteride or any 5-alpha-reductase inhibitor).
9. Females suffering from other hair loss disorders, such as alopecia areata, scarring alopecia, and telogen effluvium as determined on initial study assessment by the Investigator.
10. History of burning, flaking, itching, and stinging of the scalp.
11. History of malignancy (except SCC and BCC skin cancers) or undergoing chemotherapy or radiation treatments.
12. A known history of autoimmune thyroid disease, any other thyroid disorder/abnormality or other autoimmune disorders that are not controlled in the opinion of the investigator may interfere with the study treatment.
13. A known history of depression or bi-polar disease or any other condition that may impact the subject's participation.
14. Known history or recent blood work indicating iron deficiency, bleeding disorders or platelet dysfunction syndrome as well as subjects taking anticoagulant therapy, antiplatelet medications, more than one (1) 325 mg ASA on a daily basis or smokers with usage > 20 cigarettes/day.
15. Individuals with self-reported uncontrolled diseases (e.g., diabetes, hypertension, hyperthyroidism, hypothyroidism, etc.). All medical conditions that are under control with or without treatment will be considered on an individual basis by the Investigator.
16. Females with self-reported active hepatitis, immune deficiency, HIV or autoimmune disease.
17. Females having a known active dermatologic condition which, in the opinion of the examining Investigators, might place the subject at a greater risk or interfere with clinical evaluations (e.g., seborrheic dermatitis, psoriasis, atopic dermatitis, advanced skin cancer, etc.).
18. Use of any medications that are known to potentially cause hair loss or affect hair growth, as determined by the PI.
19. Is involved in any injury litigation claims.

    -

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 1. Females, age 40-65, who are perimenopausal, menopausal or post-menopausal. Perimenopausal is defined as increased variability in menstrual cycle length and defined as persistent difference of 7 days or more in length of consecutive cycles. Later stages include amenorrhea for 60 days or longer and/or vasomotor symptoms. These should have been present for at least 6 months prior to study. Menopause is defined as absence of menstrual bleeding for at least 12 months or 12 months status post complete Hysterectomy with Oophorectomy.
Enrollment: 70 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Terminal Hairs in the Target Area of the Scalp | 180 days
  Terminal hair is defined as coarse hair, short or long, found on the scalp with minimum cross-sectional diameter of 40 micrometers.
Number of Vellus Hairs in the Target Area of the Scalp | 180 days
  Vellus hair is defined as fine, short hairs found on the scalp with maximum cross-sectional diameter of 40 micrometers.
Number of Total Hairs in the Target Area of the Scalp | 180 days
  Total Hairs equals the sum of Terminal and Vellus Hairs in the Target Area

SECONDARY OUTCOMES:
Number of terminal hairs, number of vellus hairs, and number of total hairs in the target area of the scalp | nine (9) month and twelve (12) month visits
  Terminal hair is defined as coarse hair, short or long, found on the scalp with minimum cross-sectional diameter of 40 micrometers. Vellus hair is defined as fine, short hairs found on the scalp with maximum cross-sectional diameter of 40 micrometers. Total Hairs equals the sum of Terminal and Vellus Hairs in the Target Area
Dino-Lite microscopic photographs for terminal hair diameter measurements in the target area | Day 0, Day 90, Day 180, Day 270, Day 360
  Ten (10) terminal hairs just outside the border of the 2 cm x 2 cm area used for the Hair Check Hair Mass Index (HMI) will be randomly chosen (not all from one direct area) and cut at the surface of the scalp thus not creating any bald patches. The Dino-Lite Microscope will then be used to measure the diameter of each of the ten (10) hairs at 1mm from the cut end of the hair. All calibrations and measurement will be done at the setting of 230X. The ten (10) hair measurements will then be recorded on the Hair Diameter Log Form. All ten (10) diameters will be added together and then divided by 10 to attain an average hair diameter for the area and the average diameter will be recorded in the CRF. See Appendix IV.
Hair Washing Procedure in clinic for Hair Shedding Counts | Day 0, Day 90, Day 180, Day 270, Day 360
  Subjects will be instructed to wash their hair at home 24 hours in advance of study visits 1, 2, 3, 4 and 5. Subjects will then have their hair washed (shampooed) with a gentle shampoo in the office over a sink containing cheesecloth. The cheesecloth will be positioned to collect shedding hair. The number of hairs collected in the cheesecloth will be counted and recorded. Subjects will be allowed to dry and style their hair. Subjects will have their hair washed and shedding hairs counted on Visits 1, 2, 3, 4 and 5. See Appendix V.
Blinded Physician Global Hair Assessment for Hair Growth and Hair Quality | Day 90, Day 180, Day 270, Day 360
  The treating investigator will complete this live assessment by circling the number on the scale that corresponds to the description that best fits the current global growth improvement and current hair quality Investigator Assessment Scale
  * 3 Greatly increased
  * 2 Moderately increased
  * 1 Slightly increased 0 No change
    * 1 Slightly worsened
    * 2 Moderately worsened
    * 3 Greatly worsened
Women's Hair Loss Quality of Life Questionnaire | Day 0, Day 90, Day 180, Day 270, Day 360
  Please complete the following questions by circling the number in the column which best describes your opinion for each characteristic.
  Very Much (4) A Lot (3) A Little (2) Not At All (1) Not Relevant (0)
  1. I am embarrassed by my thinning hair.
  2. Because of my thinning hair, I avoid social gatherings.
  3. I don't like meeting new people as I feel they are judging me because of my thinning hair.
  4. I avoid going out during the day because of my thinning hair.
  5. My condition impacts my emotional state at work.
  6. I feel my thinning hair has impacted my ability to succeed in interviews.
  7. My condition has prevented my participation in a sports activity.
  8. My condition impacts my self esteem.
  9. My condition makes me feel self conscious about my thinning hair.
  10. Because of my thinning hair, I fear being the center of attention.
  11. I feel my thinning hair is affecting my personal relationships.
  12. Because of my thinning
Self-Assessment Questionnaire | Day 90, Day 180, Day 270, Day 360
  Please complete the following questions by circling the number in the column which best describes your opinion for each characteristic; from +3 (greatly increased/improved) to -3 (greatly decreased/worsened)
  Greatly Increased/Improved +3
  Moderately Increased/Improved +2
  Slightly Increased/Improved +1
  No Change 0
  Slightly Decreased/Worsened -1
  Moderately Decreased/Worsened -2
  Greatly Decreased/Worsened -3
  Overall hair growth Overall hair volume Scalp coverage Thickness of hair body Hair amount Hair quality Hair color Hair shine Hair strength Softness of hair body Amount of new hair Hair growth rate Hair length Ease of styling Overall hair appearance Sleep Quality Overall Well-Being Nail strength +3 Nail Growth rate Growth of Eyebrow hair Growth of eyelashes Skin smoothness Overall skin health Energy levels Libido (Sex drive)
  Please complete the following questions by circling the number in
Subject Treatment Satisfaction and Ease of Use Questionnaires | Day 90, Day 180, Day 270, Day 360
  Subject Treatment Satisfaction:
  Please circle the number on the scale that corresponds to the description that you believe best fits your current satisfaction with the study treatment.
  Subject Satisfaction Scale Description
  * 3 Extremely Satisfied
  * 2 Moderately Satisfied
  * 1 Slightly Satisfied 0 No change
    * 1 Slightly Unsatisfied
    * 2 Moderately Unsatisfied
    * 3 Greatly Unsatisfied
Subject Hair Satisfaction Questionnaire | Day 90, Day 180, Day 270, Day 360
  Questionnaire
  Subject Hair Satisfaction Questionnaire:
  Please check the box next to the description of your current state of hair health, which most accurately describes your current feelings of how satisfied you are with the amount and quality of hair on your scalp, including scalp coverage, volume and overall appearance.
  Subject Satisfaction Scale Description
  * 3 Extremely Satisfied
  * 2 Moderately Satisfied
  * 1 Slightly Satisfied 0 No change
    * 1 Slightly Unsatisfied
    * 2 Moderately Unsatisfied
    * 3 Greatly Unsatisfied
Menopausal Rating Scale Questionnaire | Day 0, Day 90, Day 180, Day 270, Day 360
  Questionnaire This is a standardized scale and cannot be copied into this document.

CONTACTS AND LOCATIONS:
Overall Officials: Glynis Ablon, MD, FAAD, Principal Investigator — Ablon Skin institute and Research Center
Locations (1):
- Ablon Skin Institute & Research Center, Manhattan Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ablon G, Kogan S, Raymond I. A Long-Term Study of the Safety and Efficacy of a Nutraceutical Supplement for Promoting Hair Growth in Perimenopausal, Menopausal, and Postmenopausal Women. J Drugs Dermatol. 2022 Jul 1;21(7):783. doi: 10.36849/JDD.776. PMID 35816069
- [Derived] Ablon G, Kogan S. A Randomized, Double-Blind, Placebo-Controlled Study of a Nutraceutical Supplement for Promoting Hair Growth in Perimenopausal, Menopausal, and Postmenopausal Women With Thinning Hair. J Drugs Dermatol. 2021 Jan 1;20(1):55-61. doi: 10.36849/JDD.5701. PMID 33400421